CLINICAL TRIAL: NCT01195584
Title: Minimal Access Surgical Technique (MAST) in Obese Patients in Degenerative Lumbar Disease
Status: Completed | Type: Observational
Sponsor: General Hospital Amstetten (Other)
Responsible Party: Principal Investigator, Dr. Wolfgang Senker, Principal Investigator, General Hospital Amstetten
Other Study IDs: 1-Senker
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Degenerative Lumbar Disease
Keywords: complication rate in 3 cohorts (BMI < 25, > 25 and > 30)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- BMI < 25: Body Mass Index (WHO) established by WHO. BMI < 25 has been defined as 'normal weight'.
- 25 >= BMI < 30: Body Mass Index (WHO) established by WHO. BMI >= 25 and < 30 has been defined as 'overweight'.
- BMI >= 30: Body Mass Index (WHO) established by WHO. BMI > 30 has been defined as 'obese'.

SUMMARY:
The study concerns a retrospective analysis of all subjects operated as of 1st Jan 2008 using Minimal Access Surgical Technique (MAST). The study is descriptive in nature and will present the observation of all cumulated patients operated with MAST.

The study data will include the general health information of the subjects prior to surgery, information on the surgery such as OP time, blood loss, and the postoperative wound healing process (until discharge), which is on average the 10th postoperative day.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

* all patients who underwent minimal access spinal surgery for degenerative lumbar disease fusion surgery
* patient older than 18 years
* all products have been used within intended use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent minimal access spinal surgery for degenerative lumbar disease fusion surgery.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Senker, MD, Principal Investigator — General Hospital Amstetten
Locations (1):
- General Hospital Amstetten, Amstetten, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients fulfilling in- and exclusion criteria were enrolled into the retrospecitve study. All consecutive 72 patients who signed the patient informed consent were included. Patients were stratified in three groups according to their body mass index (BMI) established by WHO. Enrollment period from January 2009 - August 2010
Groups:
- BMI < 25: Body Mass Index (BMI) according to WHO definition. BMI < 25 is defined as 'normal weight'.
- 25 <= BMI < 30: Body Mass Index (BMI) according to WHO definition. BMI >= 25 and < 30 is defined as 'overweight'.
- BMI >= 30: Body Mass Index (BMI) according to WHO definition. BMI >= 30 is defined as 'obese'.
Period: Overall Study
Arm/Group | BMI < 25 | 25 <= BMI < 30 | BMI >= 30
Started | 20 | 25 | 27
Completed | 20 | 25 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMI < 25 | 25 <= BMI < 30 | BMI >= 30 | Total
Number analyzed (Participants) | 20 | 25 | 27 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 17 | 40
  >=65 years | 6 | 16 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.1) | 67.2 (12.7) | 62.8 (11.3) | 61.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 18 | 42
  Male | 11 | 10 | 9 | 30
Region of Enrollment [Number; unit: participants]
  Austria | 20 | 25 | 27 | 72

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complications in the BMI Groups During Post Operative Hospitalization.
Description: Postoperative complications related to the operation within the body mass index groups. A complication is any harmful event occuring during the surgery until hospital discharge.
Time Frame: at hospital discharge
Population: Analysis per protocol
Measure: Number; unit: Events during hospitalization
Groups:
- Complications: Postoperative complications; complications include fever, subfebrile temerature, neurogenic deficit, temorary meningism, pulmonary embolism, TIA, cardiac ischemia, urinary tract infection, respiratory infection and pneumonia
Arm/Group | Complications
Number analyzed (Participants) | 72
Events during hospitalization
  BMI < 25 | 8
  25 >= BMI < 30 | 9
  BMI >= 30 | 20

2. Secondary Outcome: Operation Duration
Description: Duration of the operation in minutes.
Time Frame: after surgery
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Duration: Duration of surgery
Arm/Group | Duration
Number analyzed (Participants) | 72
Minutes
  BMI < 25 | 156.8 (41.6)
  25 >= BMI < 30 | 186.2 (67.8)
  BMI >= 30 | 205.4 (76.0)

3. Secondary Outcome: Blood Loss
Description: Loss of blood during surgical procedure in milliliters.
Time Frame: after surgery
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Blood Loss
Number analyzed (Participants) | 72
ml
  BMI < 25 | 165.4 (306.5)
  25 >= BMI < 30 | 284.4 (375.1)
  BMI >= 30 | 169.8 (175.0)

4. Secondary Outcome: Number of Spine Segments
Description: Number of affected spine segments. One spine segment is defined as 2 vertebral bodies and the intervertebral disc (between the 2 vertebral bodies). For this study the number fo affected spine segments is identical to the number of operated intervertebral discs.
Time Frame: peri operative
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: spine segments
Groups:
- Number of Segments: Number of affected spine segments
Arm/Group | Number of Segments
Number analyzed (Participants) | 72
spine segments
  BMI < 25 | 1.9 (0.8)
  25 >= BMI < 30 | 2.3 (1.4)
  BMI >= 30 | 2.2 (1.1)

5. Secondary Outcome: Drainage
Description: Drainage during hospitalization. The drainage was placed during the surgery and has been removed prior to hospital discharge. The amount of drainage in milliliters has been measured.
Time Frame: at hospital discharge
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Hospitalization: Days of hospitalization
Arm/Group | Hospitalization
Number analyzed (Participants) | 72
ml
  BMI < 25 | 165.6 (246.8)
  25 >= BMI < 30 | 150.4 (125.6)
  BMI >= 30 | 152.0 (141.5)

6. Secondary Outcome: Days of Hospitalization
Description: Total time of hospitalization.
Time Frame: at hospital discharge
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Hospitalization
Number analyzed (Participants) | 72
Days
  BMI < 25 | 8.4 (2.17)
  25 >= BMI < 30 | 11.2 (8.67)
  BMI >= 30 | 10.7 (3.51)

ADVERSE EVENTS:
Time Frame: Events have been recorded at hospital discharge for each patient
Description: Patients enrolled consecutively.
  Only patients who signed patient informed consent have been included. The study describes the method of minimally invasive surgery and records complications related to the operation, adverse events are not linked to medical device.
Arm/Group | BMI < 25 | 25 <= BMI < 30 | BMI >= 30
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 8/20 | 9/25 | 20/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMI < 25 (N=20) | 25 <= BMI < 30 (N=25) | BMI >= 30 (N=27)
Fever (Infections and infestations) | 3 (3) | 3 (3) | 9 (9) — Fever, defined as body temerature > 38°C
Subfebrile temperature (Infections and infestations) | 3 (3) | 6 (6) | 9 (9) — Increase in body temperature < 38°C
Neurogenic deficit (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Temporary meningism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischemic Attack (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac Ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study is retrospective and all patients during the timeframe (who signed the patient informed consent) have been included into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes